CLINICAL TRIAL: NCT07394621
Title: Kinesiophobia Affects Functional Capacity in Patients With Implanted Left Ventricular Assist Devices
Brief Title: Kinesiophobia in Patients With Implanted Left Ventricular Assist Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Rafet Umut Erdoğan, Research Assistant, Marmara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 25.01.2024/22
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Kinesiophobia (Fear of Movement)
Keywords: kinesiophobia; functional capacity; LVAD
MeSH Terms: conditions — Kinesiophobia | interventions — Walk Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Recommendation Group (Experimental): Patient who recevied physical activity recommendations after LVAD implementation
  Interventions: Diagnostic Test: Physical Activity Recommandations

INTERVENTIONS:
Diagnostic Test: Physical Activity Recommandations — Patients with implanted LVADs will be given recommendations for physical activities they can incorporate into their daily lives.
  Other Names: 30 seconds sit to stand test; 2 minute walk test

SUMMARY:
The goal of this prospective and cross-sectional observational study is to learn if the presence and changes in kinesiofobia (fear of movement) affect functional capacity levels in heart failure patients who are transplant candidates and have been implanted with a Left Ventricular Assist Device (LVAD). The main questions it aims to answer are:

i) Does the level of kinesiofobia change significantly 1 month after LVAD implantation? ii) Do changes in kinesiofobia levels predict changes in functional exercise capacity (measured by the 2-Minute Walk Test and 30-Second Sit-to-Stand Test)? Researchers will compare pre-discharge (baseline) measurements to 1-month post-discharge follow-up measurements to see if improvements in kinesiofobia correlate with improved functional mobility and endurance.

Participants will:

i) Complete the Tampa Scale of Kinesiofobia (TSK) to assess their fear of movement.

ii) Perform the 2-Minute Walk Test (2MWT) to evaluate functional exercise capacity and mobility.

iii) Perform the 30-Second Sit-to-Stand Test (30STS) to determine functional endurance and lower extremity performance.

iv) Receive standardized physical activity recommendations upon discharge. v) Return for a follow-up assessment one month later to repeat the same battery of tests.

ELIGIBILITY:
Inclusion Criteria:

* Being a heart transplant candidate and having undergone LVAD implantation,
* Having a left ventricular ejection fraction (LVEF) <30%,
* Not having developed any surgical or medical complications in the early period after implantation,
* Being referred to the study by a cardiologist at the time of discharge,
* Being able to read and write and volunteering to participate in the study.

Exclusion Criteria:

* Those with evidence of active infection following implantation,
* Psychiatric problems developing after LVAD implantation that interfere with cognitive adaptation,
* Musculoskeletal problems developing after LVAD implantation,
* Cases experiencing acute cardiac problems requiring hospitalization during follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-01-04 (Actual); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale | From enrollment to the 4 weeks after the implementation
  The Tampa Scale of Kinesiofobia (TSK) is a widely used patient-reported outcome measure designed to quantify a patient's fear of movement and fear of (re)injury. It was originally developed to assess patients with chronic low back pain, but it has since been validated for various populations. It is a 17-item questionnaire where each item is scored on a 4-point Likert scale, ranging from "strongly disagree" to "strongly agree". While cut-off values can vary by population, a score higher than 37 is often considered to represent high kinesiofobia.

SECONDARY OUTCOMES:
2-Minute Walk Test | From enrollment to the 4 weeks after the implementation
30 Seconds Sit to Stand Test (30STS) | From enrollment to the 4 weeks after the implementation

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Faculty of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No